CLINICAL TRIAL: NCT04098068
Title: Phase 2 Study of MK-3475 (Pembrolizumab) in Patients With Microsatellite Unstable (MSI) Tumors
Brief Title: Study of MK-3475 (Pembrolizumab) in Patients With Microsatellite Unstable (MSI) Tumors (Cohort D)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1365 (Cohort D); MK-3475-016 (Other: Merck); NA_00085756 (Other: JHM IRB)
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: High Tumor Mutation Burden; High TMB (Tumor Mutation Burden); MSS (Microsatellite Stable)
Keywords: Mutation load; Tumor mutation load; Mutation burden; Tumor mutation burden (TMB); Hypermutation; MSI Negative with Mutator Phenotype (High Tumor Mutation Burden); TMB (Tumor Mutation Burden)
MeSH Terms: conditions — Spinocerebellar Degenerations | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MSI (Microsatellite Unstable) Negative with Mutator Phenotype (Experimental)
  Interventions: Drug: MK-3475

INTERVENTIONS:
Drug: MK-3475 — MK-3475 (pembrolizumab) 200 mg flat dose every 21 days
  Other Names: Pembrolizumab

SUMMARY:
This study will be looking at whether MK-3475 (pembrolizumab) is effective (anti-tumor activity) and safe in patients with MSI (Microsatellite Unstable) negative cancer with a mutator phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Patients with microsatellite stable tumor and a tumor mutation burden (TMB) level measured at > 20 mutations per megabase pairs (MB)
* Have measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Adequate organ function as defined by study-specified laboratory tests
* Must use acceptable form of birth control through the study and for 28 days after final dose of study drug
* Signed informed consent form
* Willing and able to comply with study procedures
* Agree to have a biopsy of their cancer
* Patients with colon cancer must have received at least two prior cancer therapy regimens.
* Patients with other cancer types must have received at least one prior cancer therapy
* Progressive disease

Exclusion Criteria:

* Patients with uncontrolled intercurrent illness, including but not limited to ongoing or active infection, systematic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric condition that would limit compliance with study requirements.
* Patients who have had chemotherapy or biological cancer therapy within 2 weeks prior to the first dose of study drug
* Patients who have had radiation within 2 weeks prior to the first dose of study drug
* Patients who have undergone major surgery within 4 weeks of dosing of investigational agent
* Patients who have received another investigational product or investigational device within 4 weeks prior to receiving study drug
* Patients who have received any of the following concomitant therapy: Interleukin-2 (IL-2), interferon, or other non-study immunotherapy regimens, immunosuppressive agents, other investigational therapies or chronic use of systemic corticosteroids within one week prior to first dose of study drug
* Patients who have received a live vaccine within 4 weeks prior to or after any dose of MK-3475 (exception: inactivated flu vaccines)
* Patients who have received growth factors, including but not limited to granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin, etc. within 2 weeks of study drug administration
* Patient who have had prior treatment with anti-PD-1 (anti-programmed cell death protein 1), anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40, anti-CD40, or anti-CTLA-4 antibodies
* Patients with history of any autoimmune disease:inflammatory bowel disease, (including ulcerative colitis and Crohn's Disease), rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus (SLE) autoimmune vasculitis, central nervous system (CNS) or motor neuropathy considered to be of autoimmune origin.
* Patients who have known history of infection with HIV, hepatitis B, or hepatitis C
* Patients with evidence of interstitial lung disease
* Systemically active steroid use
* Patients on home oxygen
* Patients with oxygen saturation of <92% on room air by pulse oximetry
* Pregnant or lactating
* Conditions, including alcohol or drug dependence, or intercurrent illness that would affect the patient's ability to comply with study visits and procedures
* Patient with known active central nervous system metastases and/or carcinomatous meningitis.
* Patients with primary brain tumors.
* Requires any other form of systemic or localized antineoplastic therapy while on study
* Has any tissue or organ allograft
* Patients with history of allogeneic hematopoeitic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2025-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (3):
- United States (3):
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MSI (Microsatellite Unstable) Negative With Mutator Phenotype: MK-3475 (pembrolizumab): MK-3475 200 mg flat dose every 21 days
Period: Overall Study
Arm/Group | MSI (Microsatellite Unstable) Negative With Mutator Phenotype
Started | 12
Completed | 2
Not Completed | 10
Not completed — Disease Progression | 7
Not completed — Withdrawal by Subject | 2
Not completed — New Cancer Diagnosis | 1

BASELINE CHARACTERISTICS:
Arm/Group | MSI (Microsatellite Unstable) Negative With Mutator Phenotype
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Patients With MSI (Microsatellite Unstable)-Negative Solid Tumor Malignancies With a Mutator Phenotype
Description: Objective Response Rate (ORR) is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions.
Time Frame: 2 years
Population: Only 11/12 were evaluable for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | MSI (Microsatellite Unstable) Negative With Mutator Phenotype
Number analyzed (Participants) | 11
Participants | 5

2. Secondary Outcome: Overall Survival (OS)
Description: OS will be measured from date of first dose until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Time Frame: 80 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MSI (Microsatellite Unstable) Negative With Mutator Phenotype
Number analyzed (Participants) | 12
months | 41.9 [9.7 to NA] — NA means that there were an insufficient number of events to estimate the upper bound confidence interval

3. Secondary Outcome: Progression-Free Survival (PFS) in Patients Using RECIST 1.1(Response Evaluation Criteria In Solid Tumors)
Description: PFS is defined as the number of months from the date of first dose to disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MSI (Microsatellite Unstable) Negative With Mutator Phenotype
Number analyzed (Participants) | 12
months | 6.8 [2 to NA] — NA means that there were an insufficient number of events to estimate the upper bound confidence interval

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) is defined as the number of patients achieving a complete response (CR) or partial response (PR) or stable disease (SD) based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: 2 years
Population: Only 11/12 were evaluable for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | MSI (Microsatellite Unstable) Negative With Mutator Phenotype
Number analyzed (Participants) | 11
Participants | 7

5. Secondary Outcome: Number of Patients Experiencing a Grade 3 or Above Treatment-related Toxicity
Description: When calculating the incidence of AEs, each adverse event (AE) (as defined by NCI CTCAE v4.03) will be counted only once for a given subject.
Time Frame: 28 months
Measure: Count of Participants; unit: Participants
Arm/Group | MSI (Microsatellite Unstable) Negative With Mutator Phenotype
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events assessed for up to 28 months. All-Cause Mortality assessed for up to 80 months.
Arm/Group | MSI (Microsatellite Unstable) Negative With Mutator Phenotype
All-Cause Mortality (participants affected / at risk) | 4/12
Serious Adverse Events (participants affected / at risk) | 6/12
Other Adverse Events (participants affected / at risk) | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSI (Microsatellite Unstable) Negative With Mutator Phenotype (N=12)
Congestive heart failure (Cardiac disorders) | 1 (1)
Disease progression (General disorders) | 2 (2)
Opioid use disorder (Injury, poisoning and procedural complications) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diffuse large B cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSI (Microsatellite Unstable) Negative With Mutator Phenotype (N=12)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 1 (1)
Cellulitis (Immune system disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Conjunctival erythema (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
COVID infection (Infections and infestations) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (2)
Dental pain (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diabetes mellitus (Endocrine disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (6)
Dry eye (Eye disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema (General disorders) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophageal dysmotility (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 5 (7)
Fever (General disorders) | 1 (1)
Ganglion cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hernia (Injury, poisoning and procedural complications) | 1 (1)
Hyperbilirubinemia (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (3)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 3 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (4)
Nocturia (Renal and urinary disorders) | 1 (1)
Oral thrush (Infections and infestations) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Pelvic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (14)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Investigations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT04098068/Prot_SAP_000.pdf